CLINICAL TRIAL: NCT04651829
Title: Suspicion of Non IgE-mediated Cow's Milk Protein Allergy: Prevalence and Evolution
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Anaïs Lemoine, Dr, MD, Hôpital Armand Trousseau
Other Study IDs: CMPA
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Food Allergy in Infants; Proctocolitis; Atopic Dermatitis; Reflux, Gastroesophageal; Tolerance
MeSH Terms: conditions — Proctocolitis; Dermatitis, Atopic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: oral food challenge 1 — First oral food challenge after a short period of several weeks of avoidance of CMP to confirm diagnosis of CMPA
Other: oral food challenge 2 — Second oral food challenge to test tolerance after 4 months of age if confirmed CMPA

SUMMARY:
Cow's milk protein allergy (CMPA) is often evoked in infants, in particular in front of delayed symptoms such as rectal bleeding, atopic dermatitis, excessive crying, reflux, failure to thrive... But in case of non IgE-mediated CMPA, the only way to diagnose this allergy is to proceed to an elimination-reintroduction test over a period of 2 to 4 weeks, to improve symptoms first, and then provoke them. Even if the diagnosis is confirmed, we speculate that non IgE-mediated CMPA has a faster resolution than other CMPA.

The first aim of this study is to estimate the prevalence of non IgE-mediated CMPA in a cohort of infants with delayed symptoms which could be relied to a CMPA. The second goal is evaluate the age of tolerance in non IgE-mediated CMPA with oral food challenge for milk ever 2 months after 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* infants under 4 months age with delayed symptoms evoking CMPA

Exclusion Criteria:

* exclusively breastfed infants
* no improvement of symptoms despite amino acid formula
* patients with symptoms of food protein induced enterocolitis
* patients who do not have diagnostic oral food challenge within 3 months after the start of elimination diet

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants under 4 months of age consulting for delayed symptoms evoking CMPA are prospectively included. All these infants benefit from a CMP elimination diet by replacing their usual formula with an extensive CMP hydrolysate, hydrolysed rice-protein formula, or an amino acid-based formula (AAF). Only children whose symptoms disappear after this exclusion diet are selected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
prevalence of CMPA in patients with suspicion of non IgE-mediated CMPA | 2 to 8 weeks after inclusion
  We proceed to an elimination-reintroduction test of the culprit food (CMP) in patients with delayed symptoms of non IgE-mediated CMPA (rectal bleeding, atopic dermatitis, reflux, excessive crying, failure to thrive...) after a period of two to eight weeks of exclusion of CMP.
  If symptoms disappear after CMP elimination, and reappear after CMP reintroduction, the diagnosis of CMPA is confirmed.

SECONDARY OUTCOMES:
age of tolerance of confirmed non IgE-mediated CMPA | after 4 months of age, and at least after 2 months of elimination diet, and then ever 2 months until tolerance
  We proceed to an oral food challenge (OFC) for CMP every 2 months, after the age of 4 months, and after at least 2 months of elimination diet. If symptoms occur after OFC, the patient is still allergic. If no symptom occur after OFC, the patient is considered as tolerant for CMP, and that determine age of tolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric nutrition and gastroenterology department, Trousseau Hospital, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided